CLINICAL TRIAL: NCT01017627
Title: A Case Controlled Study to Determine the Impact of Adherence to Anemia Management Policy on Repeat Hospitalization in ESRD
Brief Title: Impact of Adherence to Anemia Management Policy on Repeat Hospitalization in End Stage Renal Disease (ESRD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Raymond Hakim, M.D., Ph.D., Fresenius Medical Care North America
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20090068
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Mortality
Keywords: ESRD; Anemia; Hospitalizations; Mortality
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early anemia management (Other): Upon return to the dialysis unit following hospitalization, patients will be immediately identified and have immediate implementation of the unit anemia protocol rather than waiting for the next regularly scheduled unit labs and regular follow-up. Thus, labs will be obtained within the first 3-7 days following hospitalization and appropriate titration of Epo and iron medications within the 7 days after discharge from hospital and under the direction of the pre-specified algorithm used in the patient's facility; all drug dosing will comply with package insert instructions
  Interventions: Other: Early anemia diagnosis and treatment
- case control (Other): Each case will be "data-matched" to an intra-facility (primary control), and then an inter-facility (validation control) control patient. Matching criteria will be by age, gender, diabetic status, attending nephrologist, length of hospitalization stay, and hospital discharge date (to minimize the difference in the date between the case and control). These patients did not have early intervention but followed the usual practice of waiting for the next regularly scheduled dialysis unit labs with anemia management to follow using the regular unit algorithm.
  Interventions: Other: No change from normal routine

INTERVENTIONS:
Other: Early anemia diagnosis and treatment — Patients returning to the unit are immediately assessed and treated for anemia
  Arms: Early anemia management
Other: No change from normal routine — Normal unit policy for labs and anemia treatment
  Arms: case control

SUMMARY:
The investigators hypothesize that the post-hospitalized patient status is characterized by subacute and reversible metabolic and hematological changes that, if addressed and treated in a timely manner, would result in a reduced risk for repeat hospitalization. Consequently, a structured quality improvement program, focused on increasing adherence to company wide anemia management policies (ie hemoglobin monitoring within the first 3-5 days post-hospitalization, followed by an appropriate EPO dose modification within the 7 days post-hospitalization), will significantly decrease the risk of hospital re-admission in the 30 days after discharge.

DETAILED DESCRIPTION:
The post-hospitalization quality improvement project will be piloted across 30 Fresenius clinics. Targeted enrollment of 1500 episodes of hospitalization in which the patient returns after discharge to resume outpatient dialysis.

Patient outcomes will be followed for up to 30 days from the time of discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* resumption of routine outpatient chronic hemodialysis within three days of discharge from hospital admission
* enrolled in a facility-based anemia management program

Exclusion Criteria:

* enrolled in hospice
* previous hospitalization within the past 30 days (ie. patients discharged from a repeat hospitalization)
* anticipated discharge from the outpatient dialysis facility within 30 days (ie anticipated transfer to another facility or hospice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
composite of death or repeat hospitalization within the 30 days after discharge from a previous hospitalization | one year to accumulate 1500 hospitalizations

SECONDARY OUTCOMES:
hemoglobin, transferrin saturation, albumin, white blood cell count, and C-reactive protein* levels measured in the period following hospitalization and change relative to values measured prior to hospitalization (where available). | one year to accumulate 1500 hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hakim, M.D., Ph.D., Principal Investigator — Fresenius Medical Services
Locations (42):
- United States (42):
  - Denver Central, Denver, Colorado
  - St. John's, Jacksonville, Florida
  - JAX Beach, Jacksonville, Florida
  - Prairie, Chicago, Illinois
  - Tri Counties, Decatur, Indiana
  - Huntington, Huntington, Indiana
  - Floyd County, New Albany, Indiana
  - South Louisville, Louisville, Kentucky
  - Breaux Bridge, Breaux Bridge, Louisiana
  - Delta, Delta, Louisiana
  - East Lafayette, Lafayette, Louisiana
  - Methuen, Methuen, Massachusetts
  - Roxbury, Roxbury, Massachusetts
  - Battle Creek, Battle Creek, Michigan
  - East Lansing, East Lansing, Michigan
  - Oshtemo, Kalamazoo, Michigan
  - Lansing, Lansing, Michigan
  - Saganaw Riverside, Saginaw, Michigan
  - Saginaw, Saginaw, Michigan
  - Eupora, Eupora, Mississippi
  - Meridian, Meridian, Mississippi
  - Yokna River, Oxford, Mississippi
  - Independence Centerpoint, Independence, Missouri
  - Desert Inn, Las Vegas, Nevada
  - South Pecos, Las Vegas, Nevada
  - Briggs Ave, Durham, North Carolina
  - Freedom Lake, Durham, North Carolina
  - Boardman, Boardman, Ohio
  - Cortland, Cortland, Ohio
  - Elyria, Elyria, Ohio
  - North Randall, North Randall, Ohio
  - Westlake, Westlake, Ohio
  - Willoughby, Willoughby, Ohio
  - Twin Oaks, Beaverton, Oregon
  - Clackamas, Clackamas, Oregon
  - Fresenius Medical Services, Brentwood, Tennessee
  - Smyrna, Smyrna, Tennessee
  - West Nashville, West Nashville, Tennessee
  - North Fort Worth, Fort Worth, Texas
  - Tarrant County, Fort Worth, Texas
  - Waco, Waco, Texas
  - Waco West, Waco, Texas

REFERENCES:
- [Background] Wingard RL, Pupim LB, Krishnan M, Shintani A, Ikizler TA, Hakim RM. Early intervention improves mortality and hospitalization rates in incident hemodialysis patients: RightStart program. Clin J Am Soc Nephrol. 2007 Nov;2(6):1170-5. doi: 10.2215/CJN.04261206. Epub 2007 Oct 17. PMID 17942761